CLINICAL TRIAL: NCT05327569
Title: The Efficacy of Myofascial Chain Release Techniques in Patients With Patellofemoral Pain Syndrome.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Emel Mete, research assistant, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022/0076
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-04

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Patellofemoral Pain Syndrome; Fascia; Myofascial Release Therapy
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Intervention Model Description: There will be two groups in this study. Each group will consist of 30 patients aged 25-50 years with patellofemoral pain syndrome. A total of 60 participants will take part in the study. Conventional physiotherapy will be applied to the control group, while myofascial release techniques will be applied to the experimental group in addition to conventional physiotherapy
Who Masked: Outcomes Assessor
Masking Description: Participants will be divided into two groups using block randomization method. Participants will be randomly allocated into 2 blocks of 30 participants in each group using a random number generation technique by computer. All assessments will be done by researcher who were not in the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): xperimental group will consist of 30 patients with diagnosed Patellofemoral pain syndrome, aged between 25-50 years. In addition to the conventional physiotherapy program, myofascial chain release techniques will be applied to this group.
  Myofascial release technique will be applied to the center of coordination points in the anterior superficial myofascial chain of the body. There are a total of 8 points on this myofascial chain. Pressure will be applied to each point with 6 repetitions and lasting approximately 5-6 seconds.
  Participants will be treated for a total of 6 weeks, 2 days a week. Each treatment session will last 45 minutes.
  Interventions: Other: Myofascial Chain Release Techniques
- Control group (No Intervention): Control group will consist of 30 patients with diagnosed Patellofemoral pain syndrome, aged between 25-50 years. Only conventional physiotherapy program will be applied to this group.
  Conventional treatment will consist of muscle strengthening, stretching exercises and patellar mobilization. The muscle groups to be strengthened are: M. gluteus maximus, M. gluteus medius, M. Quadriceps, Core group of muscles. The muscle groups and tendons to be stretched are: M. Hamstrings, achilles tendon and iliotibial band. The exercises will be performed as 10 repetitions and 3 sets. Participants will be treated for a total of 6 weeks, 2 days a week. Each treatment session will last 45 minutes.

INTERVENTIONS:
Other: Myofascial Chain Release Techniques — Myofascial release technique will be applied to the center of coordination points in the anterior superficial myofascial chain of the body. There are a total of 8 points on this myofascial chain. Pressure will be applied to each point with 6 repetitions and lasting approximately 5-6 seconds.
  Arms: Experimental group

SUMMARY:
The aim of this study was to evaluate the effects of myofascial release techniques applied on the superficial anterior myofascial chain of the body on pain, functional status, posture, biomechanical and viscoelastic properties of myofascial tissues in patients with patellofemoral pain syndrome.

There will be two groups in this study. Each group will consist of 30 patients aged 25-50 years with patellofemoral pain syndrome. A total of 60 participants will take part in the study. Conventional physiotherapy will be applied to the control group, while myofascial release techniques will be applied to the experimental group in addition to conventional physiotherapy. Treatment programs will be applied to both groups 2 days a week for 6 weeks. Postural problems that can be seen in the superficial anterior myofascial chain line will be evaluated. These problems: forward head, q-angle, genu varum, genu valgum, foot postural problems and pelvic tilt. In addition to all these assessments, knee pain, lower extremity functionality and biomechanical properties of the anterior myofascial tissue will be evaluated.

DETAILED DESCRIPTION:
Many factors such as lower extremity malalignment, quadriceps muscle weakness, hamstring, gastrocnemius, tensor fascia latae muscle shortness, iliotibial band tension, lower extremity malalignment have been shown to be effective in the development of Patellofemoral pain syndrome. But it has been reported in recent studies that myofascial problems can be related with patellofemoral pain syndrom. It is stated that the fascial chain containing the Patellofemoral pain syndrome-related regions is the Superficial Anterior Chain, and this chain starts from the toe extensors and ends at the masteoid process. The aim of this study was to evaluate the effects of myofascial release techniques applied on the superficial anterior myofascial chain of the body on pain, functional status, posture, biomechanical and viscoelastic properties of myofascial tissues in patients with patellofemoral pain syndrome.

There will be two groups in this study. Each group will consist of 30 patients aged 25-50 years with patellofemoral pain syndrome. A total of 60 participants will take part in the study. Conventional physiotherapy will be applied to the control group, while myofascial release techniques will be applied to the experimental group in addition to conventional physiotherapy. Treatment programs will be applied to both groups 2 days a week for 6 weeks. Postural problems that can be seen in the superficial anterior myofascial chain line will be evaluated. These problems: forward head, q-angle, genu varum, genu valgum, foot postural problems and pelvic tilt. In addition to all these assessments, knee pain, lower extremity functionality and biomechanical properties of the anterior myofascial tissue will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Patellofemoral pain syndrome,
* Volunteers between the ages of 25-50,
* Having pain in the retropatellar region for at least 6 months that is not a result of trauma,
* Not having received medical treatment and/or physiotherapy for PFPS in the last 6 months.

Exclusion Criteria:

* Having history of lower extremity, pelvis and spine surgery/fracture in the last 6 months,
* Having orthopedic (Anterior cruciate ligament rupture, Meniscal tears, etc), neurological (Multiple sclerosis, paralysis-paralysis, etc.) and/or rheumatological (rheumatoid arthritis, ankylosing spondolitis, etc.) problems,
* Pregnancy ,
* Having a history of connective tissue disease,
* Using sedatives and/or muscle relaxants that may alter muscle tone.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-20 (Estimated); Primary Completion 2023-05-02 (Estimated); Study Completion 2023-06-10 (Estimated)

PRIMARY OUTCOMES:
Knee pain | Change from baseline knee pain at week 6.
  Visual Analogue Scale will be used in the assessment of pain severity. It expresses pain severity between a score of 0 (no pain) and 10 (unbearably severe pain).
Forward head | Change from baseline craniovertebral angle at week 6.
  The craniovertebral angle will be considered in determining the forward tilt of the head. In this study, markers will be placed on the mastoid process and C7 spinous process to determine the craniovertebral angle. Photographs of the participants will be taken from the front and side, and then the craniovertebral angle will be calculated using the Tracker 4.11.0 software on these photos. Forward head posture is characterized as pathologic when the craniovertebral angle (CVA) is ≥50°.
Q-Angle | Change from baseline Q-angle at week 6.
  For the Q angle, the angle between a straight line from the SIAS to the center of the patella and the line from the center of the patella to the center of the tuberositas tibia will be measured with a goniometer. While the Q angle can be between 6° and 27°, its approximate average value is 15°. Increasing or decreasing the Q angle increases the pressure in the lateral and medial compartments of the patellofemoral joint.
Genu varum | Change from baseline genu varum at week 6.
  The individual in the standing position is asked to unite the lower extremities while maintaining 0° extension of the knees. The distance between the medial condyles is measured as the medial malleolar are in contact. If the distance is more than 1 cm, it indicates the genu varum.
Genu Valgum | Change from baseline genu valgum at week 6.
  The individual in the standing position is asked to unite the lower extremities while maintaining 0° extension of the knees. The distance between the medial malleolar is measured as the medial condyles are in contact. If the distance is more than 1 cm, it indicates the genu valgum.
Pes planus | Change from baseline pes planus at week 6.
  Pes Planus will be evaluated with navicular drop test. The distance between the navicular bone and the ground is measured while the individual sits on the chair with the hip-knee joint in 90º flexion and the subtalar joint in neutral position. Then, the distance between the navicular bone and the ground is measured again while the individual is standing in a position with equal weight on both extremities. The difference between the two measurements is recorded. 10 mm or more difference is considered pes planus.
Foot posture | Change from baseline foot posture at week 6.
  Foot posture will be evaluated using the Foot posture index, a six item foot posture assessment tool, where each item is scored between -2 and +2 to give a sum total between -12 (highly supinated) and +12 (highly pronated). Items include: talar head palpation, curves above and below the lateral malleoli, calcaneal angle, talonavicular bulge, medial longitudinal arch, and forefoot to rearfoot alignment.
Pelvic tilt | Change from baseline pelvic tilt at week 6.
  The position of the pelvis will be evaluated with a digital pelvic inclinometer device to determine whether the pelvis has tilted anteriorly or posteriorly. The digital pelvic inclinometer is a valid and reliable method for the evaluation of pelvic tilt. The device consists of two calipers and the calipers are placed on the SIAS (spina illaca anterior posterior) and SIPS (spina illaca posterior superior) of the pelvis. The score on the digital display is recorded. "-" values indicate posterior pelvic tilt, "+" values indicate anterior pelvic tilt.
Lower extremity functionality | Change from baseline lower extremity functionality at week 6.
  Lower extremity functional scale will be used. This scale is a valid and reliable scale used in musculoskeletal problems affecting the lower extremities. It consists of 20 items. Each item is scored between 0-4. The total score is between 0-80. Higher scores indicate better functional status.
elacticity | Change from baseline Biomechanical and viscoelastic properties of myofascial tissues at week 6.
  Elacticity of myofascial tissues will be evaluated with MyotonPro digital palpation device which is a valid and reliable. In the measurements, the Myoton probe will be placed perpendicular to the fibers of the tissue to be measured and when the probe reaches a sufficient depth, 3 repetitive mechanical stimulus (15ms, 0.40N) will be given to the tissue that has pre-compressed (0.18N). Measurements were taken 3 times from each point and the average values will be used in statistical analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Emel Mete, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No